CLINICAL TRIAL: NCT06521931
Title: A Single-arm, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamics and Immunogenicity of PN20 for the Prevention of Chemotherapy-induced Thrombocytopenia in Patients With Lymphoma or Solid Tumor
Brief Title: A Study of PN20 for the Prevention of Chemotherapy-induced Thrombocytopenia in Lymphoma or Solid Tumor Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Peg-Bio Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CQPJ-PN20-Ib
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PN20 group (Experimental): thrombopoietin receptor agonist
  Interventions: Drug: PN20

INTERVENTIONS:
Drug: PN20 — Three dose cohorts: 0.2, 0.5 and 0.75 mg/kg, subcutaneous injections, on Day 1 of chemotherapy cycle before the administration of chemotherapy drugs

SUMMARY:
The main aim of this clinical trial is to assess the safety and tolerability of PN20 in adult patients with chemotherapy-induced thrombocytopenia (CID). The main questions it aims to answer are:

* Is PN20 safe in these patients?
* Could these patients potentially benefit from PN20 prevention? Participants will
* Receive subcutaneous injections of PN20 according to weight on the first day of chemotherapy cycle, within 1 hour before the administration of chemotherapy drugs,
* Visit the clinic on Day 1 (D1), D2, D3, D4, D5, D8, D11, D13, D15 and D21 for assessment.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label, dose escalation study to evaluate the safety, tolerability, pharmacokinetic, pharmacodynamics and immunogenicity of PN20 for the Prevention of Chemotherapy-induced Thrombocytopenia in Adult Patients With Lymphoma or Solid Tumor.

This study was divided into two phase, single-dose and multiple-dose. After single-dose period (21 days), if the subject meets the multiple-dose criteria, he or she can enter the multiple-dose phase for the second cycle of PN20 prevention. Subjects could receive a maximum of two cycles of PN20 prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years, regardless of gender;
2. Diagnosed with lymphoma or solid tumor by pathological histology or cytology examination;
3. Currently receiving a 21-day chemotherapy regimen, using one or more of the following or similar drugs: gemcitabine; platinums, including carboplatin, nedaplatin, cisplatin, lobaplatin, etc.; anthracyclines, including doxorubicin, daunorubicin, epirubicin, etc.; taxanes, including paclitaxel, docetaxel, etc.; alkylating agents, including cyclophosphamide, ifosfamide, etc.;
4. The current chemotherapy regimen should be consistent with that of the previous chemotherapy cycle before enrollment, including the type and dosage of the drugs, and no medication or dosage adjustments are allowed;
5. Platelet count (PLT) was between 75 and 150×10^9/L (including the critical value) one day before the start of chemotherapy in the first treatment cycle or before enrollment;
6. There was a decrease in PLT to 25×10^9/L≤ PLT <75×10^9/L during the previous chemotherapy cycle before enrollment;
7. Expected survival ≥ 12 weeks;
8. Eastern Cooperative Oncology Group (ECOG) Physical Score is ≤ 2;
9. No fertility plan during the trial and within 6 months after the end of the follow-up, and agree to take medically recognized contraceptive measures (such as complete abstinence, condoms, contraceptive rings, ligation, drug contraception, etc.) to avoid pregnancy for themselves or their partners;
10. Be able to understand the requirements and procedures of the protocol, voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. With thrombocytopenia caused by non-chemotherapy within 6 months before screening, including but not limited to ethylenediaminetetraacetic acid (EDTA)-dependent pseudothrombocytopenia, hypersplenism, infection and bleeding;
2. With other hematopoietic diseases other than lymphoma and chemotherapy induced thrombocytopenia, including leukemia, primary immune thrombocytopenia, myeloproliferative diseases, multiple myeloma and myelodysplastic syndrome;
3. The tumor has already undergone bone marrow invasion or metastasis;
4. With active central nervous system metastasis (such as clinical symptoms, cerebral edema, requiring hormone intervention (excluding maintenance of low-dose hormones)), progression of brain metastasis, and carcinomatous meningitis. Subjects with previously treated brain metastases who meet the following conditions may participate in the study: clinical stability has been maintained for ≥ 2 months, and systemic hormone therapy (prednisone or other equivalent doses of hormones at a dose of >10 mg/day) has been discontinued for >4 weeks;
5. Acute or active bleeding of clinical significance (such as gastrointestinal or central nervous system) within 7 days before screening;
6. Have a history of any arteriovenous thrombosis within 6 months before screening;
7. Have a history of major cardiovascular disease within 6 months before screening (such as congestive heart failure (New York Heart Association (NYHA) heart function score III-IV), arrhythmias known to increase the risk of thromboembolic events (atrial fibrillation, etc.), coronary stent implantation, angioplasty or coronary artery bypass grafting);
8. Accompanying diseases that the investigator believes the investigational drug may cause unnecessary risks of, such as: severe cardiovascular and cerebrovascular diseases, digestive system diseases, liver and kidney dysfunction diseases, or a family history of mental illness;
9. Laboratory examination abnormalities during the screening period (baseline), such as:

   1. Blood biochemistry: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin ≥ 3 times the upper limit of normal (ULN) (if liver metastasis exists, ALT, AST, total bilirubin can be ≥ 5 × ULN); serum creatinine ≥ 1.5 × ULN;
   2. Blood routine: absolute neutrophil value <1.5×10^9/L; hemoglobin < 80 g/L;
10. Abnormal electrocardiogram of clinical significance during screening or prolonged QT/QTc interval, such as QTcF ≥ 450ms (male) or 470ms (female); family history of QT prolongation;
11. Active hepatitis B (hepatitis B virus titer > 1,000 copies/ml or 200IU/ml); hepatitis C virus infection (HCV-RNA Above the detection limit); preventive antiviral treatment other than interferon is allowed. For patients with hepatocellular carcinoma (HCC), hepatitis B virus titer> 10,000 copies/ml or 2000IU/ml; human immunodeficiency virus antibody (HIV), syphilis positive;
12. Received platelet transfusion within 5 days before the first dose;
13. Anticoagulants (heparin, warfarin, apixaban, bivalirudin, etc.), antiplatelet drugs (clopidogrel, aspirin, etc.), fibrinolytic drugs (urokinase, etc.) were used for prevention or treatment within 1 week before the first dose;
14. Received other drugs with platelet-raising effects (e.g., caffeic acid tablets, leucogen tablets, aminopeptide tablets, or platelet-raising capsules, etc.) within 1 week before the first dose; received recombinant human thrombopoietin (rh-TPO) or used recombinant human interleukin-11 (rhIL-11), thrombopoietin receptor agonist (TPO-RA) within 10 days before the first dose or 5 half-lives of the drug (whichever is longer);
15. Currently receiving or received radiotherapy within 3 months before screening;
16. Received bone marrow transplantation or stem cell infusion within 1 year before screening;
17. Allergic to the investigational drug or excipients (such as histidine, glycine, mannitol, sucrose) or previously experienced life-threatening systemic allergic reaction;
18. Used other clinical trial drugs or devices within 4 weeks before the first dose;
19. Other conditions the investigator believes would be unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
AE in single-dose phase | Day 1-21 of Cycle 1 (each cycle is 21 days)
  The incidence of adverse events related to PN20 within 21 days after a single dose
The proportion of patients with PLT ≥ 100×10^9/L in multiple-dose phase | Day 21 of Cycle 2 (each cycle is 21 days)
  The proportion of subjects whose platelet count (PLT) reached ≥ 100 × 10^9/L at the end of the second chemotherapy cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital
Locations (6):
- China (6):
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Yiyang Central Hospital, Yiyang, Hunan
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan